CLINICAL TRIAL: NCT01163773
Title: Milk Consumption and the Metabolic Syndrome in Menopausal Women
Acronym: MILK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Dairy Farmers of Canada (Other)
Responsible Party: Benoît Lamarche, PhD, Institute of Nutraceutical and Functional Foods (INAF), Laval University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: INAF-2004-039
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Milk; Metabolic syndrome; Blood lipids; Menopausal women
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MILK — Consumption of the 2 experimental diets
  1. Milk diet
  2. Control diet

SUMMARY:
Cardiovascular disease (CVD) represents the first cause of mortality in industrialized countries such as Canada and the United States. In that regard, it is being increasingly recognized that a significant proportion of CVD events may be attributable to the presence of a cluster of metabolic and physiological perturbations defined as the metabolic syndrome (MetS). The National Cholesterol Education Program- Adult Treatment Panel III (NCEP-ATP III) has recently proposed a clinical definition to identify individuals with the MetS. This definition is based on the presence of at least three of the following five characteristics: 1- abdominal obesity, 2- hypertriglyceridemia, 3- reduced plasma HDL-C levels, 4- high blood pressure, 5- high fasting blood glucose levels. Recent data have suggested that the MetS based on this definition was associated with a 2 to 5 fold increase in the risk of CVD in men as well as in women. These are alarming figures since it has been suggested that as much as 35 to 45% of female aged > 65 years in the US may have the MetS. It is therefore imperative to develop new preventive strategies that will be efficacious in attenuating the impact of the MetS on the progressing rates of CVD in women. In that context, there is accumulating evidence to suggest that milk and dairy products may beneficially modify several components of the MetS. However, most of the available data to date are based on observational studies or interventional studies with minimal nutritional control. Thus, metabolically controlled studies that document the impact of milk consumption on cardiovascular risk factors associated with the MetS in women defined a priori as having the MetS are utterly lacking.

The purpose of this study was to investigate the impact of milk consumption on features of the MetS in menopausal women presenting one or more features of the MetS.

DETAILED DESCRIPTION:
The proposed research will be undertaken as a randomized, cross-over, nutritionally controlled study, with participants being subjected to two 6-week isocaloric diets separated by a 4-week washout period. No stratification was considered since the population recruited will be relatively homogeneous. The experimental diet (designed as 'Milk') will be formulated so that the percentage of daily calories from fat (30%), saturated fat (10%), carbohydrates (55%) and proteins (15%) will conform to most of the dietary recommendations of the American Heart Association and the NCEP for primary prevention of CVD, with the exception of saturated fats (slight excess) and fibers (slight deficit). The cholesterol content of the experimental diet will not exceed 200 mg/day. The only source of dairy products during the experimental phase will be from 2% fat milk. We have chosen to use 2% fat milk because this is the most frequently consumed dairy product in Canada. Two percent fat milk also goes through minimal processing compared to milk or to other dairy products such as yogurt and cheese. Thus, bioactive components in milk are more likely to be retained in the 2% fat milk than in other more extensively processed products. The energy intake from milk will represent 20% of the consumed kcal/day. Based on a reasonable 2000 kcal/day regimen, a 20% intake attributable to 2% fat milk will correspond to 400 day/kcal, which will be derived from a 'daily dose' of 3 portions of milk/day. This dose has been shown to be effective in previous uncontrolled studies. The Control diet will be virtually identical in terms of menus, calories and macronutrient composition, with the exception that milk will be formally excluded from the regimen. The energy intake and changes in macronutrient composition attributable to the milk component in the experimental diet will be compensated in the control diet by modifying the protein, carbohydrate and lipid component of the various recipes.

A 4-week stabilization run-in period will precede the randomization of participants. During this run-in period, participants will be asked and instructed to comply to the NCEP-ATP III prudent diet. They will be asked to maintain their body weight constant during this period. Milk consumption will be adapted during this period to comply to the recommendations of NCEP-ATP III. The washout period between the two experimental diets will last 4 weeks and will also consist of NCEP-ATP III recommended diet. It must be stressed that foods will not be provided during the run-in and wash-out periods. These periods are imposed to minimize the inter- and intra-individual variability before and between the experimental phases.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women (absence of menses > 12 months and FSH > 40 IU/ml), aged between 45 and 65 years
* Presenting 1 or more features of the MetS based on the NCEP-ATP III definition
* Average consumption of milk/dairy products fewer than 2 portions/d (≤ 1.9)
* Stable body weight (+/- 2 kg) for 6 months before the beginning of the study

Exclusion Criteria:

* Previous history of cardiovascular disease, type 2 diabetes and monogenic dyslipidemia
* Subjects taking medications for hyperlipidemia, hypertension or hormonal replacement therapy
* Endocrine disorders
* Smoking
* Food allergies, milk aversion or intolerant to lactose
* Women with extreme nutritional habits such as vegetarism or alcohol consumption > 2 drinks/day

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Plasma TG levels (MetS criteria) | At the beginning and the end of the two 6-week diets
HDL-C levels (MetS criteria) | At the beginning and the end of the two 6-week diets
Systolic and diastolic blood pressure (MetS criteria) | At the beginning and the end of the two 6-week diets
Fasting blood glucose (MetS criteria) | At the beginning and the end of the two 6-week diets

SECONDARY OUTCOMES:
Anthropometric measures (waist and hip circumferences) | At the beginning and the end of the two 6-week diets
LDL and HDL particle size | At the beginning and the end of the two 6-week diets
Markers of the oxidative stress (i.e. oxLDL and 8-iso-PGF2a levels) | At the beginning and the end of the two 6-week diets
Markers of a pro-inflammatory state (i.e. C-reactive protein and IL-6 levels) | At the beginning and the end of the two 6-week diets
Surrogates of cholesterol absorption and synthesis | At the beginning and the end of the two 6-week diets

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Institute of Nutraceutical and Functional Foods (INAF), Laval University
Locations (1):
- Institute of Nutraceutical and Functional Foods (INAF), Laval University, Québec, Quebec, Canada